CLINICAL TRIAL: NCT06036368
Title: 6-weeks, Open-label, Single-Site Study to Evaluate Safety, Tolerability and Efficacy of the Home-based Peroneal Electrical Transcutaneous NeuroModulation (Peroneal eTNM®) Treatment Via Nerve Stimulator URIS ITM in Treatment of Symptoms Related to Movement Disorders in Subjects With Parkinson's Disease (PD) and Essential Tremor (ET)
Brief Title: Study to Evaluate Safety and Efficacy of Peroneal Transcutaneous NeuroModulation in Subjects With Parkinson's Disease and Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stimvia s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS004-PD
Record Dates: First submitted 2023-08-18; First posted 2023-09-13 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease; Essential Tremor
Keywords: Parkinson's Disease (PD) and Essential Tremor (ET); Peroneal Electrical Transcutaneous NeuroModulation
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peroneal eTNM arm (Experimental): All patients will receive treatment with peroneal eTNM
  Interventions: Device: Peroneal electrical transcutaneous neuromodulation (peroneal eTNM®)

INTERVENTIONS:
Device: Peroneal electrical transcutaneous neuromodulation (peroneal eTNM®) — This is a non-invasive intervention, which utilizes direct trancutaneous, electrical stimulation of the peroneal nerve

SUMMARY:
This is a 6-week exploratory clinical study, designed to test whether treatment with peroneal electrical trans-cutaneous stimulation can have a beneficial effects on symptoms associated with Parkinson's diseases and essential tremor.

DETAILED DESCRIPTION:
This is a 6-week, open-label, single site clinical study designed to test whether treatment with peroneal electrical trans-cutaneous stimulation (eTNM) can have a beneficial effects on symptoms associated with Parkinson's diseases (PD) and essential tremor (ET). Eligible patients will be treated with eTNM at home for 6 weeks. Primary endpoint in this study is tolerability and safety, secondary and exploratory endpoints are various scale designed to capture improvements in the most bothersome symptoms of PD or ET.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Competent and willing to provide written, informed consent to participate in the study
* Stable dose of any chronic medications, if applicable, for 30 days prior to study entry
* Willing to comply with study protocol requirements
* Subject agrees not to participate in another study from 30 days prior the screening visit until the final study visit
* For subjects with PD:

Bradykinesia in "on" period based on clinical assessment Rigidity in "on" period based on clinical assessment Hand/arm exhibiting tremor (resting and/or intentional and/or postural) ≥ grade 1 as assessed by the MDS-UPDRS tremor score in "on" period

• For subjects with ET: Visible hand/arm and/or foot/leg tremor (resting and/or intentional and/or postural) ≥ grade 1 as assessed by the TETRAS

Exclusion Criteria:

* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator
* Suspected or diagnosed epilepsy or other seizure disorder
* Severe degree of disability or dependence in daily activities >grade 3 as measured by modified Rankin Scale (mRS)
* Presence of clinical signs or diagnosis of dementia
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* Presence of clinical signs of peripheral neuropathy on lower limbs
* Presence of chorea and/or dyskinesia
* Clinical symptoms or diagnosis of major depressive disorder
* Presence of any other neurodegenerative disease. These may include multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Botulinum toxin injection within 6 months prior to study enrollment
* Participation in another interventional clinical trial in the last 30 days, which may confound the results of this study, unless approved by the Sponsor
* Subject is breastfeeding, pregnant, intends to become pregnant during the study, or of childbearing potential, sexually active and not practicing a highly reliable method of birth control (these are methods with a failure quotient of <1% year such as hormonal implants, injectable contraceptives, oral contraceptives of combination type, intra-uterine pessaries restricted to hormone contraceptive coil, sexual abstinence or vasectomy of the partner). The pregnancy test in urine at both Visits 1 and 2 needs to be negative in women of childbearing potential.
* Subjects unable to communicate effectively with the investigator and staff
* Life expectancy less than 6 months
* Subject with active malignant disease
* Subject with alcohol (more than 100 mg ethanol per day) or drug abuse during the recruitment and during the trial course
* Subject who, in the opinion of the physician, may interfere with optimal participation in the clinical trial or may pose a risk to the subject
* Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Baseline to end of treatment at 6 weeks
  Incidence of treatment emergent adverse events

SECONDARY OUTCOMES:
Response of the condition on the therapy | Baseline to end of treatment at 6 weeks
  Change in Patient Global Impression of Improvement scale (Scores 1-7, lower number = better)

OTHER OUTCOMES:
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  The Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score (both total score and subscores) (applicable only for subjects with PD)(0-260, lower score = better)
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Essential tremor rating assessment scale (TETRAS) score (applicable only for subjects with ET, 0-64, lower scores = better))
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Bradykinesis and rigidity measured by Five Times Sit to Stand Test (FTSTS) (applicable only for subjects with PD, time in seconds, lower = better))
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Bradykinesis and rigidity measured objectively using the 10 meter Walking Speed Test (WST) (time in seconds, lower = better)(applicable only for subjects with PD)
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Effect on patient's daily activities measured by Bain and Findley Activities of Daily Living (BF-ADL) (25-100, lower score = better)
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Degree of disability measured by modified Rankin Scale (mRS) (0-6, lower score= better)
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Quality of life measured by European Quality of Life-5 Dimensions questionnaire (EQ-5D-5L)(0.532-1.000, higher score = better)
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Disease-specific quality of life measured by Parkinson's Disease Questionnaire (PDQ -39)(0-100, lower score = better)
Exploratory efficacy | Baseline to end of treatment at 6 weeks
  Patient's satisfaction using Treatment Satisfaction Visual Analog scale (TS-VAS)(0-100, higher score = better)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, MD, PhD, Principal Investigator — Cerebrovaskulární poradna s.r.o., Ostrava
Locations (1):
- Cerebrovaskulární poradna s.r.o., Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: No